CLINICAL TRIAL: NCT02812992
Title: A Multicenter Phase 4 Geriatric Assessment Directed Trial to Evaluate Gemcitabine +/- Nab-paclitaxel in Elderly Pancreatic Cancer Patients
Brief Title: Geriatric Assessment Directed Trial to Evaluate Gemcitabine +/- Nab-paclitaxel in Elderly Pancreatic Cancer Patients
Acronym: GrantPax
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-GER-0115
Record Dates: First submitted 2016-06-07; First posted 2016-06-24 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Adenocarcinoma Pancreas
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GO-GO arm (Active Comparator): Nab-paclitaxel 125 mg/m^2 i.v. over 30 minutes followed by gemcitabine infusion 1000 mg/m^2 on days D1, D8, D15 of a 28-day cycle.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- SLOW-GO arm (Active Comparator): Gemcitabine 1000 mg/m^2 i.v. on days D1, D8, D15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine
- FRAIL arm (Active Comparator): Best supportive care as determined by the investigator.
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: Nab-paclitaxel
  Other Names: Abraxane®
  Arms: GO-GO arm
Drug: Gemcitabine
  Arms: GO-GO arm; SLOW-GO arm
Other: Best Supportive Care
  Arms: FRAIL arm

SUMMARY:
The GrantPax study is a multicenter phase 4 geriatric assessment directed trial to evaluate gemcitabine +/- nab-paclitaxel in elderly pancreatic cancer patients. The primary objective is that CGA-stratified patients do not decline in their CGA performance in response to chemotherapy measured as a loss of five points or less in the Barthel's ADL, (ADL1 vs. ADL2 during core CGA assessment).

DETAILED DESCRIPTION:
The hypothesis of the proposed study is that individualized assessment directed treatment algorithms identifies elderly patients, who benefit from combined nab-paclitaxel/gemcitabine therapy. The project uses a CGA, which includes various tests and scoring systems, to stratify patients as "GO-GO", "SLOW-GO" or "FRAIL" patients. Depending on test results patients receive chemotherapy (GO-GO group: nab-paclitaxel/gemcitabine; SLOW-GO group: gemcitabine monotherapy) or best supportive care (FRAIL group). After the first cycle of chemotherapy (4 weeks) a subsequent CGA and a safety assessment will be performed to assign patients to their definite treatment arm. The primary objective is that CGA-stratified patients do not decline in their CGA performance in response to chemotherapy measured as a loss of five points or less in the Barthel's ADL (ADL1 vs. ADL2 during core CGA assessment).

ELIGIBILITY:
Inclusion Criteria 1 - Chemotherapy arms (Go-Go, Slow-Go):

1. Patients ≥ 70 years of age.
2. Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas.
3. At least one measurable lesion of disease according to RECIST 1.1 criteria.
4. No prior chemotherapy (except fluoruracil or gemcitabine in an adjuvant setting at least > 6 months prior enrollment).
5. Adequate end organ function:

   * renal function: serum creatinine ≤ 1.5 x ULN or GFR ≥ 30mL/min.
   * hematopoietic function: white blood cell (WBC) count ≥3000/μL, absolute neutrophil count (ANC) ≥ 1500/μL, platelets ≥10^5/μL, hemoglobin level >9.0 g/dL
   * liver function: total bilirubin ≤1.5 x ULN, AST / ALT ≤3.0 x ULN
6. Cooperation and willingness to complete all aspects of the study
7. Written informed consent to participate in the study

Inclusion criteria 2 - FRAIL arm:

1. Patients ≥ 70 years of age.
2. Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas.
3. No prior chemotherapy (except fluoruracil or gemcitabine in an adjuvant setting at least > 6 months prior enrollment).
4. Cooperation and willingness to complete all aspects of the study
5. Written informed consent to participate in the study

Exclusion Criteria 1 - Chemotherapy arms (Go-Go, Slow-Go):

1. Patients <70 years of age.
2. Papillary cancer, cholangiocellular carcinoma, neuro-endocrine tumors.
3. Patient has a severe and/or uncontrolled medical disease (i.e. uncontrolled active infection, uncontrolled hypertension/ diabetes or cardiac disease).
4. Patient has received any other investigational product within 28 days prior study entry.
5. Patient is < 5 years free of another primary malignancy (except: not currently clinically significant nor requiring active intervention)
6. Hypersensitivity against gemcitabine or nab-paclitaxel.
7. Major surgery ≤ 28 days prior to study entry.
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
9. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
10. Any other chemotherapy at start.
11. Any psychiatric illness that would affect the patient's ability to understand the demands of the clinical trial.
12. Parallel participation in another clinical trial or participation in another clinical trial within the last 30 days or 7 half-lifes of a study medication, whichever is of longer duration, prior study start.
13. Patient has already been recruited in this trial.
14. Patients who do not understand the nature, the scope and the consequences of the clinical trial.
15. Patient who might be dependent on the sponsor, the study site or the investigator.
16. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 Nr. 4 AMG.

Exclusion criteria 2 - FRAIL arm:

1. Patients <70 years of age.
2. Papillary cancer, cholangiocellular carcinoma, neuro-endocrine tumors.
3. Patient has received any other investigational product within 28 days prior study entry.
4. Patient is < 5 years free of another primary malignancy (except: not currently clinically significant nor requiring active intervention)
5. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
6. Any chemotherapy at study start.
7. Any psychiatric illness that would affect the patient's ability to understand the demands of the clinical trial.
8. Parallel participation in another clinical trial or participation in another clinical trial within the last 30 days or 7 half-lifes of a study medication, whichever is of longer duration, prior study start.
9. Patient has already been recruited in this trial.
10. Patients who do not understand the nature, the scope and the consequences of the clinical trial.
11. Patient who might be dependent on the sponsor, the study site or the investigator.
12. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 Nr. 4 AMG.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Barthel's ADL [Barthel's scale in activities of daily living] | 4 weeks
  Loss of five points or less in the Activity of Daily Living (Barthel's ADL; assessed during 2nd CGA) after first cycle of chemotherapy (or after 4 weeks in BSC group) compared to the initial ADL for each treatment groups.

SECONDARY OUTCOMES:
CGA [Comprehensive Geriatric Assessment] | 4 weeks
  Scores before and after 1st treatment cycle (CGA1+2 further CGA scores 3+4 - if available) or after 28 days of BSC
ECOG [Eastern Cooperative Oncology Group] | 4 weeks
  Scores before and after 1st treatment cycle (CGA1+2 further CGA scores 3+4 - if available) or after 28 days of BSC
ADL (Barthel) [Activities of Daily Living] | 4 weeks
  Scores before and after 1st treatment cycle (CGA1+2 further CGA scores 3+4 - if available) or after 28 days of BSC
IADL (Lawton/Browdy) [Instrumental Activities of Daily Living] | 4 weeks
  Scores before and after 1st treatment cycle (CGA1+2 further CGA scores 3+4 - if available) or after 28 days of BSC
G8-Questionnaire | 4 weeks
  Scores before and after 1st treatment cycle (CGA1+2 further CGA scores 3+4 - if available) or after 28 days of BSC
CR [Complete Response] | 12 months
PR [Partial Response] | 12 months
DCR [Disease Control Rate] | 12 months
ORR [Objective Response Rate] | 12 months
AEs/SAEs [Adverse Events/Serious Adverse Events] | 12 months
PFS [Progression Free Survival] | 12 months
OS [Overall Survival] | 12 months
Percentage of patients receiving at least one chemotherapy in each treatment group | 12 months
Percentage of patients escalating treatment | 12 months
Duration of treatment | 12 months
Cumulative dose | 12 months
QoL [Quality of Life] | 12 months
  time to QoL deterioration [loss of 10 points or more in QLQ-C30]
Discrepancy between CGA strata estimation by the investigator and true CGA assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Ebert, Prof., Principal Investigator — Universitätsklinikum II. Medizinische Klinik
Locations (1):
- Universitätsklinikum Mannheim II. Medizinische Klinik, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Betge J, Chi-Kern J, Schulte N, Belle S, Gutting T, Burgermeister E, Jesenofsky R, Maenz M, Wedding U, Ebert MP, Haertel N. A multicenter phase 4 geriatric assessment directed trial to evaluate gemcitabine +/- nab-paclitaxel in elderly pancreatic cancer patients (GrantPax). BMC Cancer. 2018 Jul 18;18(1):747. doi: 10.1186/s12885-018-4665-2. PMID 30021548